CLINICAL TRIAL: NCT02854930
Title: Near Death Experience (NDE) and Migraine
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-47
Record Dates: First submitted 2016-08-01; First posted 2016-08-04 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Migraine; Near Death Experience
Keywords: Clinical death; state of consciousness
MeSH Terms: conditions — Migraine Disorders; Death

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: questioning

SUMMARY:
Migraine is a common disabling primary headache disorder. Epidemiological studies have documented its high prevalence and high socio-economic and personal impacts. Migraine affects more than 20% of the French population. However, the physiopathology of migraine is always partially known. Cortical spreading depression (CSD) is the widely accepted as the electrophysiologic substrate of migraine aura. CSD is a slowly propagating wave of transient neuronal and glial depolarization. The near death experience (NDE) is a rare, but well known phenomenon. NDE are profound psychic experiences commonly occuring in life-threatening conditions. Among the neurological hypotheses, epilepsy, temporal lobe disorders , REM-sleep intrusion have been discussed. However, the role of DCE has never been discussed. The goals of this study are : to see if there is an epidemiological link between NDE and migraine/ to specify if NDE was followed by a migrainous headache.

ELIGIBILITY:
Inclusion Criteria:

* Subject who experienced an NDE defined by the occurrence, when the subject is in a state of clinical death or a particular state of consciousness of a following event: body output experience, disembodiment, for a tunnel and / or light;
* Topic recorded in the EMI database (Dr. Postel, National Center for Education, Research and Information on the conscience;
* Topic agreeing to participate in the study.

Exclusion Criteria:

* Patient mental condition or disorder or psychiatric history or any other factor limiting the ability to participate in an informed manner and compliant to the study;
* Other than obtained Participation Agreement.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: subject who experienced a near death experience (NDE).
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-01 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Quality of life | one day

CONTACTS AND LOCATIONS:
Overall Officials: Urielle Desalbres, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille Hôpital de la Timone, Marseille, France